CLINICAL TRIAL: NCT04622592
Title: A Randomized, Partially-Blinded, Active Comparator-Controlled, Dose-Ranging, Safety, Tolerability, and Immunogenicity Phase 1/2 Study of an Adjuvanted Seasonal Recombinant Quadrivalent VLP Influenza Vaccine in Adults 65 Years of Age and Older
Brief Title: Adjuvanted Seasonal Recombinant Quadrivalent Virus-Like Particles (QVLP) Influenza Vaccine in Adults 65 Years of Age and Older
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CP-PRO-AdjQVLP-020
Record Dates: First submitted 2020-10-16; First posted 2020-11-10 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Influenza
Keywords: vaccine; safety; immunogenicity; plant-made; virus-like particle; hemagglutinin
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- QVLP15+Full AS03 (Experimental): Participants received one intramuscular (IM) injection (total volume 0.7 mL) of 15 μg/strain of the Quadrivalent virus-like particle (VLP) Influenza Vaccine adjuvanted with full dose of AS03 on Day 0 into the deltoid region of the non-dominant arm (if possible).
  Interventions: Biological: Instramuscular vaccine
- QVLP15+Half AS03 (Experimental): Participants received one IM injection (total volume 0.7 mL) of 15 μg/strain of the Quadrivalent VLP Influenza Vaccine adjuvanted with half dose of AS03 on Day 0 into the deltoid region of the non-dominant arm (if possible).
  Interventions: Biological: Instramuscular vaccine
- QVLP30+Full AS03 (Experimental): Participants received one IM injection (total volume 0.7 mL) of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine adjuvanted with full dose of AS03 on Day 0into the deltoid region of the non-dominant arm (if possible).
  Interventions: Biological: Instramuscular vaccine
- QVLP30+Half AS03 (Experimental): Participants received one IM injection (total volume 0.7 mL) of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine adjuvanted with half dose of AS03 on Day 0 into the deltoid region of the non-dominant arm (if possible).
  Interventions: Biological: Instramuscular vaccine
- QVLP45+Full AS03 (Experimental): Participants received one IM injection (total volume 0.7 mL) of 45 μg/strain of the Quadrivalent VLP Influenza Vaccine adjuvanted with full dose of AS03 on Day 0 into the deltoid region of the non-dominant arm (if possible).
  Interventions: Biological: Instramuscular vaccine
- QVLP45+Half AS03 (Experimental): Participants received one IM injection (total volume 0.7 mL) of 45 μg/strain of the Quadrivalent VLP Influenza Vaccine adjuvanted with half dose of AS03 on Day 0 into the deltoid region of the non-dominant arm (if possible).
  Interventions: Biological: Instramuscular vaccine
- QVLP30 unadjuvanted (Active Comparator): Participants received one IM injection of 0.7 mL of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine unadjuvanted on Day 0 into the deltoid region of the non-dominant arm (if possible).
  Interventions: Biological: Instramuscular vaccine
- Fluzone HD Quad (Active Comparator): Participants received one IM injection of 0.7 mL of 60 μg/strain of the Fluzone high dose (HD) Quadrivalent Influenza Vaccine on Day 0 into the deltoid region of the non-dominant arm (if possible).
  Interventions: Biological: Instramuscular vaccine

INTERVENTIONS:
Biological: Instramuscular vaccine — On Day 0, a single injection of the assigned dose of the vaccine into the deltoid region of the arm

SUMMARY:
This randomized, partially-blinded, active comparator-controlled was conducted at multiple sites globally. The composition of QVLP used in this study includes a mix of recombinant H1, H3, and two B hemagglutinin proteins expressed as VLPs and is based on the 2020-2021 influenza virus strains.

In this study, 3 dose levels (15 μg/strain, 30 μg/strain, and 45 μg/strain) of QVLP were planned to be tested in combination with 2 dose levels of AS03 adjuvant (full and half dose) in a single-dose regimen to select a dose level of QVLP and adjuvant dose level-combination that is safe and effective for further development.

Participants participated in this study for up to approximately 13 months, during which the first visit was scheduled for screening (up to 7 days in advance of vaccine administration) and the second visit on Day 0 was scheduled for vaccine administration. Telephone contacts were made on Day 1, Day 8, and monthly (starting after Day 28) until the end of the study for safety assessments, including concomitant medication use review. Blood draws at the clinic site for key safety assessments were made on Day 3, and Day 28 and for key immunogenicity assessments on Day 0, Day 28, Day 182 (6-month follow-up), and Day 365 (12-month follow-up).

DETAILED DESCRIPTION:
In this study, a partially-blinded design was applied whereby the following individuals did not have access to treatment allocation (i.e. remained "blind") throughout the entire study duration: the participants, the Investigators and all personnel involved in the clinical conduct of the study (except the staff involved in the preparation and administration of the study vaccine, the quality assurance auditor, and quality control reviewers), Medicago clinical staff and medical staff involved in safety evaluations (e.g. causality assessments), and all personnel involved in sample analysis at the central and testing laboratories.

A total of 209 participants were randomized to the study, divided into 8 groups receiving different adjuvant dose level-combinations of QVLP or Fluzone HD Quad (60 µg/strain). The majority of participants (126 participants) received QVLP 30 μg/strain with full dose AS03 (42 participants), QVLP 30 μg/strain unadjuvanted (41 participants) or Fluzone HD Quad (43 participants), while in 5 other groups with 83 participants enrolled in total the enrollment was discontinued prematurely due to recruitment challenges caused by COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Participants read, understood, and signed the informed consent form prior to participating in the study; participants also completed study-related procedures and communicated with the study staff at visits and by phone during the study;
2. Male and female participants 65 years of age and older at the Vaccination visit (Visit 2);
3. Participants had a body mass index (BMI) < 30 kg/m2 at the Vaccination visit (Visit 2);
4. Participants were considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study;
5. Participants were non-institutionalized (e.g. not living in rehabilitation centers or old-age homes; living in an elderly community was acceptable) and had no acute or evolving medical problems prior to study participation and no clinically relevant abnormalities that could jeopardize participant safety or interfere with study assessments, as assessed by the Investigator and determined by medical history, physical examination, serology, clinical chemistry and hematology tests, urinalysis, and vital signs. Investigator discretion was permitted with this inclusion criterion;

Note: Participants with a pre-existing chronic disease were allowed to participate if the disease was stable and, according to the Investigator's judgment, the condition was unlikely to confound the results of the study or pose additional risk to the participant by participating in the study. Stable disease was generally defined as no new onset or exacerbation of pre-existing chronic disease 3 months prior to vaccination. Based on the Investigator's judgment, participants with more recent stabilization of a disease were also eligible.

Exclusion Criteria:

1. According to the Investigator's opinion, significant acute or chronic, uncontrolled medical or neuropsychiatric illness. Acute disease was defined as presence of any moderate or severe acute illness with or without a fever within 48 hours prior to the Vaccination visit (Visit 2). "Uncontrolled" was defined as:

   * Requiring a new medical or surgical treatment during the 3 months prior to study vaccine administration;
   * Required any significant change in a chronic medication (i.e. drug, dose, frequency) during the 3 months prior to study vaccine administration due to uncontrolled symptoms or drug toxicity unless the innocuous nature of the medication change met the criteria outlined in inclusion criterion #5 and was appropriately justified and documented by the Investigator. Note: Investigator discretion was permitted with this exclusion criterion.
2. Any confirmed or suspected current immunosuppressive condition or immunodeficiency, including cancer, human immunodeficiency virus, hepatitis B or C infection (participants with a history of cured hepatitis B or C infection without any signs of immunodeficiency at present time were allowed). Investigator discretion was permitted with this exclusion criterion;
3. Current autoimmune disease requiring systemic treatment (such as rheumatoid arthritis, systemic lupus erythematosus, or multiple sclerosis). Investigator discretion was permitted with this exclusion criterion, and participants were eligible to participate with appropriate written justification in the source document (i.e. participants with a history of autoimmune disease who were disease-free without treatment for 3 years or more, or on stable thyroid replacement therapy, mild psoriasis [i.e. a small number of minor plaques requiring no systemic treatment], etc.);
4. Administration of any non-influenza vaccine within 30 days prior to the Vaccination visit (Visit 2); planned administration of any vaccine up to Day 28 of the study. Immunization on an emergency basis during the study was evaluated on case-by-case basis by the Investigator.

   Note: Administration of an authorized COVID-19 vaccine prior to or during the study was acceptable;
5. Administration of influenza vaccine within 6 months prior to the Vaccination visit (Visit 2) or planned administration of influenza vaccine (other than the study vaccine) up to completion of the study;
6. Administration of any adjuvanted or investigational influenza vaccine within 1 year prior to randomization or planned administration prior to the completion of the study;
7. Use of any investigational or non-registered product within 30 days or five half-lives, whichever is longer, prior to the Vaccination visit (Visit 2) or planned use during the study period. Participants who were in a prolonged post-administration observation period of another investigational or marketed drug clinical study, for which there was no ongoing exposure to the investigational or marketed product and all scheduled on-site visits were completed, were allowed to take part in this study, if all other eligibility criteria were met;
8. Administration of any medication or treatment that may alter the vaccine immune responses, such as:

   * Systemic glucocorticoids at a dose exceeding 10 mg of prednisone (or equivalent) per day for more than 7 consecutive days or for 10 or more days in total, within 1 month prior to the Vaccination visit (Visit 2). Inhaled, nasal, intraarticular, ophthalmic, dermatological, and other topical glucocorticoids were permitted;
   * Cytotoxic, antineoplastic or immunosuppressant drugs - within 36 months prior to the Vaccination visit (Visit 2);
   * Any immunoglobulin preparations or blood products, blood transfusion - within 6 months prior to the Vaccination visit (Visit 2);
9. Use of any prescription antiviral drugs with the intention of COVID-19 prophylaxis, including those that were thought to be effective for prevention of COVID-19 but had not been licensed for this indication, within 1 month prior to the Vaccination visit (Visit 2);
10. Participants at high risk of contracting SARS-CoV-2/COVID-19 infection, including, but not limited to, individuals with known close contact with:

    * anyone residing in, visiting, or working at a health care or long-term care institution (i.e. long-term care facilities, acute care hospitals, rehabilitation hospitals, mental health hospitals, emergency departments);
    * anyone with laboratory-confirmed SARS-CoV-2/COVID-19 infection within 2 weeks prior to vaccine administration;
    * anyone who traveled outside the country for any duration within 30 days before the study vaccination;
11. History of allergy to any of the constituents of QVLP, any components of Fluzone HD Quad, the adjuvant AS03, egg, or tobacco;
12. History of anaphylactic allergic reactions to plants or plants components (including fruits and nuts);
13. Participants with a history of Guillain-Barré Syndrome;
14. Personal or family (first-degree relatives) history of narcolepsy;
15. Use of prophylactic medications (e.g. antihistamines [H1 receptor antagonists], nonsteroidal anti-inflammatory drugs [NSAIDs], systemic and topical glucocorticoids, non-opioid and opioid analgesics) within 24 hours prior to the Vaccination visit (Visit 2) to prevent or pre-empt symptoms due to vaccination;
16. Had a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at the injection site that could interfere with injection site reaction rating. Investigator discretion was permitted with this exclusion criterion;
17. Participants identified as an Investigator or employee of the Investigator or clinical site with direct involvement in this study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in this study, or any employees of Medicago.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 209 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Medicago
Locations (14):
- United States (14):
  - Optimal Sites, Huntsville, Alabama
  - Synexus, Chandler, Arizona
  - Optimal Sites, San Diego, California
  - Optimal Sites, Melbourne, Florida
  - Global AES, Orlando, Florida
  - Global AES, The Villages, Florida
  - Optimal Sites, Peoria, Illinois
  - Synexus, Evansville, Indiana
  - Optimal Sites, Rockville, Maryland
  - Vitalink Research, Anderson, South Carolina
  - Vitalink Research, Columbia, South Carolina
  - Vitalink Research, Gaffney, South Carolina
  - Vitalink Research, Union, South Carolina
  - Optimal Sites, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at an equal ratio into 8 treatment groups to receive Quadrivalent Virus-Like Particles (QVLP) vaccine adjuvanted with AS03 (full and half dose), QVLP vaccine unadjuvanted or Fluzone HD Quad vaccine.
Pre-assignment Details: Participants were healthy adult males and females 65 years of age and older.
Period: Overall Study
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Started | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Vaccinated | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Completed | 18 | 9 | 38 | 16 | 21 | 13 | 38 | 36
Not Completed | 1 | 0 | 4 | 3 | 2 | 0 | 3 | 7
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 4
Not completed — Other than specified above | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Ser (SAS) was defined as all participants who received either the adjuvanted QVLP or the active comparators.
Groups:
- QVLP15+Full AS03: Participants received one IM injection (total volume 0.7 mL) of 15 μg/strain of the Quadrivalent VLP Influenza Vaccine adjuvanted with full dose of AS03 on Day 0 into the deltoid region of the non-dominant arm (if possible).
- Fluzone HD Quad: Participants received one IM injection of 0.7 mL of 60 μg/strain of the Fluzone HD Quadrivalent Influenza Vaccine on Day 0 into the deltoid region of the non-dominant arm (if possible).
- Total: Total of all reporting groups
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad | Total
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43 | 209
Age, Customized [Count of Participants; unit: Participants]
  65-74 years | 14 | 7 | 33 | 14 | 17 | 10 | 33 | 34 | 162
  ≥75 years | 5 | 2 | 9 | 5 | 6 | 3 | 8 | 9 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 24 | 10 | 10 | 4 | 24 | 29 | 115
  Male | 11 | 3 | 18 | 9 | 13 | 9 | 17 | 14 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 0 | 0 | 0 | 4 | 1 | 10
  Not Hispanic or Latino | 16 | 9 | 40 | 19 | 23 | 13 | 37 | 42 | 199
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 8
  White | 17 | 8 | 40 | 18 | 19 | 13 | 39 | 42 | 196
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunization History [Count of Participants; unit: Participants]
  Both Influenza and Non-influenza | 1 | 0 | 9 | 0 | 0 | 0 | 5 | 8 | 23
  Only influenza | 6 | 3 | 16 | 6 | 9 | 4 | 15 | 15 | 74
  Only non-influenza | 2 | 1 | 2 | 0 | 1 | 1 | 3 | 2 | 12
  None | 10 | 5 | 15 | 13 | 13 | 8 | 18 | 18 | 100

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HI) Antibody Response for Each Homologous Influenza Strain on Day 0
Description: The GMTs in each treatment group were measured using an HI assay for the homologous influenza strains: A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination)
Population: Per protocol (PP) set included participants with a Day 0 and any post-vaccination immunogenicity assessment who completed the study with no major protocol deviations related to participant eligibility, the ability to develop a valid immune response, prohibited medication use, or the immunogenicity analyses; and who received QVLP or the active comparators.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 38 | 19 | 21 | 13 | 37 | 39
titers
  H1N1 | 87.5704 [54.8902 to 139.7076] | 71.2385 [36.1378 to 140.4323] | 69.1840 [49.7233 to 96.2612] | 60.7941 [38.1065 to 96.9894] | 65.5830 [42.0562 to 102.2709] | 52.1449 [29.6458 to 91.7193] | 80.6590 [57.7141 to 112.72] | 71.9561 [51.9366 to 99.692]
  H3N2 | 42.9963 [22.1910 to 83.3079] | 35.6256 [13.6267 to 93.1394] | 53.5390 [33.5390 to 85.4653] | 28.2789 [14.5951 to 54.7919] | 26.8632 [14.3194 to 50.3954] | 57.9959 [26.0689 to 129.0241] | 53.9648 [33.5942 to 86.6876] | 50.3624 [31.7401 to 79.9107]
  B/Yamagata lineage | 27.2713 [14.0420 to 52.9642] | 58.7285 [22.3868 to 154.0659] | 35.1259 [21.9677 to 56.1656] | 24.8494 [12.7950 to 48.2607] | 23.9640 [12.7454 to 45.0573] | 21.0585 [9.4388 to 46.9827] | 31.8921 [19.8200 to 51.3171] | 31.1646 [19.6087 to 49.5307]
  B/Victoria lineage | 32.6846 [18.1258 to 58.9372] | 38.5215 [16.3560 to 90.7256] | 46.6653 [30.7568 to 70.8021] | 21.1180 [11.7113 to 38.0803] | 36.7938 [21.0003 to 64.4648] | 61.2554 [30.0331 to 124.9366] | 36.3962 [23.8547 to 55.5314] | 26.5681 [17.6053 to 40.0937]

2. Primary Outcome: GMTs of HI Antibody Response for Each Homologous Influenza Strain on Day 28
Description: as for outcome 1
Time Frame: Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
titers
  H1N1 | 296.2330 [179.6681 to 488.4226] | 419.3985 [206.7820 to 850.6303] | 222.1740 [157.4823 to 313.4401] | 168.9548 [103.8485 to 274.8785] | 174.3779 [108.5108 to 280.2268] | 214.6073 [119.1544 to 386.5261] | 165.0534 [114.7138 to 237.4834] | 208.8559 [148.7010 to 293.3456]
  H3N2 | 205.4037 [109.7143 to 384.5505] | 217.8171 [89.7300 to 528.7448] | 399.5021 [259.4647 to 615.1201] | 319.7171 [173.6539 to 588.6365] | 255.5949 [140.9883 to 463.3632] | 355.9261 [170.1736 to 744.4362] | 369.0050 [233.8149 to 582.3613] | 352.6912 [230.3416 to 540.0285]
  B/Yamagata lineage | 95.0432 [52.2252 to 172.9667] | 117.6911 [50.4649 to 274.4718] | 108.9616 [72.1607 to 164.5304] | 48.0076 [26.8043 to 85.9836] | 67.2848 [38.1259 to 118.7446] | 58.0067 [28.6740 to 117.3459] | 59.0477 [38.1940 to 91.2874] | 137.4894 [91.5389 to 206.5059]
  B/Victoria lineage | 91.4846 [53.7284 to 155.7729] | 76.9675 [36.2594 to 163.3783] | 121.7513 [84.4092 to 175.6135] | 81.3894 [48.4830 to 136.6302] | 81.3375 [49.0918 to 134.7638] | 113.1054 [60.4641 to 211.5776] | 67.2196 [45.6367 to 99.0097] | 114.1339 [79.5030 to 163.8498]

3. Primary Outcome: Percentage of Participants With Seroconversion Measured by HI Antibody Response for Each Homologous Influenza Strain on Day 28
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥4-fold increase in reciprocal HI titers between Day 0 and Day 28 or a rise of undetectable HI titer (i.e. < 10) pre-vaccination (Day 0) to an HI titer of ≥ 40 on Day 28 was measured using an HI assay for the homologous influenza strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
percentage of participants
  H1N1 | 38.9 [17.30 to 64.25] | 55.6 [21.20 to 86.30] | 36.8 [21.81 to 54.01] | 42.1 [20.25 to 66.50] | 25.0 [8.66 to 49.10] | 30.8 [9.09 to 61.43] | 29.4 [15.10 to 47.48] | 38.5 [23.36 to 55.38]
  H3N2 | 38.9 [17.30 to 64.25] | 55.6 [21.20 to 86.30] | 65.8 [48.65 to 80.37] | 63.2 [38.36 to 83.71] | 70.0 [45.72 to 88.11] | 61.5 [31.58 to 86.14] | 47.1 [29.78 to 64.87] | 64.1 [47.18 to 78.80]
  B/Yamagata lineage | 33.3 [13.34 to 59.01] | 22.2 [2.81 to 60.01] | 31.6 [17.50 to 48.65] | 21.1 [6.05 to 45.57] | 30.0 [11.89 to 54.28] | 30.8 [9.09 to 61.43] | 14.7 [4.95 to 31.06] | 38.5 [23.36 to 55.38]
  B/Victoria lineage | 44.4 [21.53 to 69.24] | 33.3 [7.49 to 70.07] | 26.3 [13.40 to 43.10] | 36.8 [16.29 to 61.64] | 30.0 [11.89 to 54.28] | 15.4 [1.92 to 45.45] | 23.5 [10.75 to 41.17] | 46.2 [30.09 to 62.82]

4. Primary Outcome: Percentage of Participants With Seroprotection Measured by HI Antibody Response for Each Homologous Influenza Strain on Day 28
Description: Seroprotection rate: the percentage of participants in a given treatment group attaining a reciprocal HI titer of ≥40 on Day 28 (the percentage of vaccine recipients with a serum HI titer of at least 1:40 following vaccination) for the homologous influenza strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
percentage of participants
  H1N1 | 100 [81.47 to 100.00] | 100 [66.37 to 100.00] | 100 [90.75 to 100.00] | 94.7 [73.97 to 99.87] | 90.0 [68.30 to 98.77] | 100 [75.29 to 100.00] | 100 [89.72 to 100.00] | 100 [90.97 to 100.00]
  H3N2 | 88.9 [65.29 to 98.62] | 88.9 [51.75 to 99.72] | 97.4 [86.19 to 99.93] | 94.7 [73.97 to 99.87] | 100 [83.16 to 100.00] | 100 [75.29 to 100.00] | 97.1 [84.67 to 99.93] | 92.3 [79.13 to 98.38]
  B/Yamagata lineage | 77.8 [52.36 to 93.59] | 88.9 [51.75 to 99.72] | 76.3 [59.76 to 88.56] | 63.2 [38.36 to 83.71] | 80.0 [56.34 to 94.27] | 76.9 [46.19 to 94.96] | 67.6 [49.47 to 82.61] | 89.7 [75.78 to 97.13]
  B/Victoria lineage | 88.9 [65.29 to 98.62] | 77.8 [39.99 to 97.19] | 97.4 [86.19 to 99.93] | 68.4 [43.45 to 87.42] | 80.0 [56.34 to 94.27] | 84.6 [54.55 to 98.08] | 82.4 [65.47 to 93.24] | 89.7 [75.78 to 97.13]

5. Primary Outcome: Geometric Mean Fold Rise (GMFR) Measured by HI Antibody Response for Each Homologous Influenza Strain (Day 28/Day 0)
Description: GMFR, the geometric mean of the ratio of GMTs (Day 28/Day 0) in each treatment group was measured using an HI assay for the homologous strains: A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination), Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
ratio
  H1N1 | 4.0142 [2.5134 to 6.4112] | 5.9788 [3.0859 to 11.5835] | 3.2024 [2.3211 to 4.4183] | 2.5570 [1.6213 to 4.0326] | 2.5408 [1.6304 to 3.9597] | 3.4414 [1.9819 to 5.9757] | 2.3058 [1.6405 to 3.2410] | 2.9661 [2.1587 to 4.0755]
  H3N2 | 4.7572 [2.6074 to 8.6794] | 5.1509 [2.2007 to 12.0561] | 8.4563 [5.5885 to 12.7956] | 8.0508 [4.4716 to 14.4949] | 6.3791 [3.5973 to 11.3124] | 7.3718 [3.6320 to 14.9624] | 7.6527 [4.9365 to 11.8637] | 7.5907 [5.0451 to 11.4208]
  B/Yamagata lineage | 3.3872 [2.1090 to 5.4401] | 2.7245 [1.3900 to 5.3402] | 3.3189 [2.3950 to 4.5993] | 1.7591 [1.1090 to 2.7904] | 2.5016 [1.5953 to 3.9227] | 2.3219 [1.3284 to 4.0586] | 1.8422 [1.3051 to 2.6005] | 4.4642 [3.2361 to 6.1584]
  B/Victoria lineage | 2.7180 [1.7465 to 4.2299] | 2.0988 [1.1229 to 3.9228] | 3.0230 [2.2264 to 4.1046] | 2.9769 [1.9293 to 4.5934] | 2.2729 [1.4941 to 3.4576] | 2.4588 [1.4564 to 4.1511] | 1.8734 [1.3579 to 2.5846] | 3.7317 [2.7594 to 5.0465]

6. Primary Outcome: Number of Participants With at Least One Immediate Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. Immediate AEs were defined as any solicited (local and systemic) and unsolicited AEs that started up to 30 minutes after vaccination. Solicited local AEs included erythema, swelling, and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck.
Time Frame: Up to 30 minutes post-vaccination
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 1 | 0 | 4 | 3 | 5 | 1 | 5 | 4

7. Primary Outcome: Number of Participants With at Least One Immediate AE of Grade 1, 2, 3, or 4
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. Immediate AEs were defined as any solicited (local and systemic) and unsolicited AEs that started up to 30 minutes after vaccination. Solicited local AEs included erythema, swelling, and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck. The intensity of the AEs was graded according to the United States Food and Drug Administration Toxicity Grading Scale: mild (Grade 1), moderate (Grade 2), severe (Grade 3), or potentially life threatening (Grade 4).
Time Frame: Up to 30 minutes post-vaccination
Population: Participants in SAS with at least one immediate AE.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 1 | 0 | 4 | 3 | 5 | 1 | 5 | 4
Participants
  Immediate solicited AE Grade 1 | 1 | 0 | 4 | 3 | 4 | 1 | 4 | 4
  Immediate solicited AE Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Immediate solicited AE Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Immediate solicited AE Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With at Least One Immediate AE Related to Vaccination
Description: An AE is defined in OM #6. Immediate AEs were defined as any solicited (local and systemic) and unsolicited AEs that started up to 30 minutes after vaccination. Solicited local AEs included erythema, swelling and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck. A related AE is an event where the investigator determined that the relationship to study vaccine was "Possibly Related", "Probably Related" or "Definitely Related". If a participant reported multiple occurrences of the same AE, only the most closely related occurrence was presented. The causal relationship of all solicited local and systemic AEs was considered related to vaccination. Participants with any related AE was reported.
Time Frame: 30 minutes post-vaccination
Population: Participants in SAS with at least one immediate AE.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 1 | 0 | 4 | 3 | 5 | 1 | 5 | 4
Participants
  Related immediate solicited AE | 1 | 0 | 4 | 3 | 5 | 1 | 5 | 4
  Related immediate unsolicited AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With at Least One Solicited Local or Systemic AE From Day 0 up to Day 7
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. Solicited local AEs included erythema, swelling, and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck.
Time Frame: Day 0 (pre-vaccination) up to Day 7
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 12 | 5 | 37 | 12 | 14 | 8 | 26 | 25

10. Primary Outcome: Number of Participants With at Least One Solicited Local or Systemic AE of Grade 1, 2, 3, or 4 From Day 0 up to Day 7
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. Solicited local AEs included erythema, swelling and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck. The intensity of the AEs was graded according to the FDA Toxicity Grading Scale: mild (Grade 1), moderate (Grade 2), severe (Grade 3), or potentially life threatening (Grade 4).
Time Frame: Day 0 (pre-vaccination) up to Day 7
Population: Participants in SAS with at least one solicited local or systemic AE.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 12 | 5 | 37 | 12 | 14 | 8 | 26 | 25
Participants
  Solicited AE of Grade 1 | 8 | 3 | 21 | 8 | 5 | 7 | 16 | 16
  Solicited AE of Grade 2 | 3 | 2 | 13 | 4 | 7 | 1 | 7 | 5
  Solicited AE of Grade 3 | 0 | 0 | 3 | 0 | 1 | 0 | 3 | 4
  Solicited AE of Grade 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With at Least One Unsolicited AE From Day 0 up to Day 28
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 6 | 4 | 6 | 3 | 1 | 0 | 8 | 7

12. Primary Outcome: Number of Participants With at Least One Unsolicited AE of Grade 1, 2, 3, or 4 From Day 0 up to Day 28
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. The intensity of the AEs was graded according to the FDA Toxicity Grading Scale: mild (Grade 1), moderate (Grade 2), severe (Grade 3), or potentially life threatening (Grade 4).
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: Participants in SAS with at least one unsolicited AE.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 1 | 0 | 8 | 7
Participants
  Unsolicited AE Grade 1 | 3 | 1 | 1 | 3 | 0 | 0 | 4 | 2
  Unsolicited AE Grade 2 | 1 | 0 | 4 | 0 | 1 | 0 | 4 | 4
  Unsolicited AE Grade 3 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 1
  Unsolicited AE Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With at Least One Unsolicited AE Related to Vaccination From Day 0 up to Day 28
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. A related AE was an event where the Investigator determined that the relationship to study vaccine was "Possibly Related", "Probably Related" or "Definitely Related". If a participant reported multiple occurrences of the same AE, only the most closely related occurrence was presented. Participants with any related AE were reported.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: Participants in SAS with at least one unsolicited AE.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 1 | 0 | 8 | 7
Participants | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 1

14. Primary Outcome: Number of Participants With at Least One Serious Adverse Events (SAE) From Day 1 up to Day 28
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. An SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event.
Time Frame: Day 1 up to Day 28
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With at Least One AE Leading to Withdrawal From the Study From Day 1 up to Day 28
Description: as for outcome 11
Time Frame: Day 1 up to Day 28
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Number of Participants With at Least One Adverse Event of Special Interest (AESI) From Day 1 up to Day 28
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. AESIs included hypersensitivity reactions, narcolepsy, Potential Immune-Mediated Diseases (pIMDs), and other AESIs. Participants with any AESI were reported.
Time Frame: Day 1 up to Day 28
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With at Least One Medically Attended AE (MAAE) From Day 1 up to Day 28
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. MAAEs are defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a healthcare provider.
Time Frame: Day 1 up to Day 28
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 2 | 0 | 3 | 1 | 1 | 0 | 7 | 7

18. Primary Outcome: Number of Participants With at Least One New Onset Clinical Disease (NOCD) From Day 1 up to Day 28
Description: All NOCDs that may plausibly have an allergic, autoimmune or inflammatory component were assessed and reported. Plausibility was interpreted broadly; the only clear exceptions were degenerative conditions such as osteoarthritis, age-related physiologic changes and life-style diseases. In this context, most cancers, cardiac conditions, and kidney diseases had to be reported.
Time Frame: Day 1 up to Day 28
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Participants With the Occurrence of Death From Day 1 up to Day 28
Description: The number of participants in each treatment group with an occurrence of death was assessed.
Time Frame: Day 1 up to Day 28
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: Number of Participants With at Least One SAE From Day 29 up to Day 182
Description: as for outcome 14
Time Frame: Day 29 up to Day 182
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 5

21. Primary Outcome: Number of Participants With at Least One AE Leading to Withdrawal From the Study From Day 29 up to Day 182
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. The number of participants with at least one AE leading to withdrawal was assessed.
Time Frame: Day 29 up to Day 182
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: Number of Participants With at Least One AESI From Day 29 up to Day 182
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. AESIs included hypersensitivity reactions, narcolepsy, pIMDs, and other AESIs. Participants with any AESI were reported.
Time Frame: Day 29 up to Day 182
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Primary Outcome: Number of Participants With at Least One MAAE From Day 29 up to Day 182
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. MAAEs are defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider.
Time Frame: Day 29 up to Day 182
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 3 | 1 | 14 | 3 | 2 | 2 | 6 | 12

24. Primary Outcome: Number of Participants With at Least One New NOCD From Day 29 up to Day 182
Description: All NOCDs that may plausibly have an allergic, autoimmune or inflammatory component were assessed and reported. Plausibility was interpreted broadly; the only clear exceptions were degenerative conditions such as osteoarthritis, age-related physiologic changes and life-style diseases. In this context, most cancers, cardiac conditions, and kidney diseases were reported.
Time Frame: Day 29 up to Day 182
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0

25. Primary Outcome: Number of Participants With an Occurrence of Death From Day 29 up to Day 182
Description: The number of participants in each treatment group with an occurrence of death was assessed.
Time Frame: Day 29 up to Day 182
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Primary Outcome: Number of Participants With at Least One SAE From Day 183 up to Day 365
Description: as for outcome 14
Time Frame: Day 183 up to the end of study (Day 365)
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 1 | 6 | 1 | 0 | 0 | 1 | 2

27. Primary Outcome: Number of Participants With at Least One AE Leading to Withdrawal From the Study From Day 183 up to Day 365
Description: as for outcome 21
Time Frame: Day 183 up to the end of study (Day 365)
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

28. Primary Outcome: Number of Participants With at Least One AESI From Day 183 up to Day 365
Description: as for outcome 22
Time Frame: Day 183 up to the end of study (Day 365)
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Primary Outcome: Number of Participants With at Least One MAAE From Day 183 up to Day 365
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. MAAEs were defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider.
Time Frame: Day 183 up to the end of study (Day 365)
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 3 | 2 | 8 | 4 | 0 | 3 | 5 | 4

30. Primary Outcome: Number of Participants With at Least One NOCD From Day 183 up to Day 365
Description: All NOCDs that may plausibly have an allergic, autoimmune or inflammatory component were assessed and reported. Plausibility should be interpreted broadly; the only clear exceptions are degenerative conditions such as osteoarthritis, age-related physiologic changes and life-style diseases. In this context, most cancers, cardiac conditions, and kidney diseases should be reported.
Time Frame: Day 183 up to the end of study (Day 365)
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0

31. Primary Outcome: Number of Participants With an Occurrence of Death From Day 183 up to Day 365
Description: The number of participants in each treatment group with an occurrence of death was assessed.
Time Frame: Day 183 up to the end of study (Day 365)
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

32. Primary Outcome: Number of Participants With Clinically Significant Abnormal Urine, Hematological, and Blood Biochemistry Values on Day 0
Description: Participants were monitored for any abnormal findings in urine parameters (urine color, glucose, occult blood, protein, specific gravity, specimen appearance, pH), hematological parameters (basophils, leukocytes, eosinophils, erythrocytes mean corpuscular hemoglobin, erythrocytes, hematocrit, hemoglobin, lymphocytes, mean platelet volume, monocytes, neutrophils, platelets), and blood chemistry parameters (alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, calcium, chloride, cholesterol, creatinine, gamma glutamyl transferase, glucose, HDL and LDL cholesterol, phosphate, potassium, protein, sodium, triglycerides, urea nitrogen). Any laboratory result outside of the testing laboratory's normal range was classified as "clinically significant" or "not clinically significant" by the site investigator, with appropriate documentation.
Time Frame: Day 0 (pre-vaccination)
Population: SAS. Only participants with at least one clinically significant laboratory parameter are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

33. Primary Outcome: Number of Participants With Clinically Significant Abnormal Urine, Hematological, and Blood Biochemistry Values on Day 3
Description: as for outcome 32
Time Frame: Day 3
Population: SAS. Only participants with at least one clinically significant abnormal laboratory finding are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants
  Urine glucose - abnormal, clinically significant | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urine occult blood - abnormal, clinically significant | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine protein - abnormal, clinically significant | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine specimen appearance - abnormal, clinically significant | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

34. Primary Outcome: Number of Participants With Clinically Significant Abnormal Urine, Hematological, and Blood Biochemistry Values on Day 28
Description: Participants were monitored for any abnormal findings in urine parameters (urine color, glucose, occult blood, protein, specific gravity, specimen appearance, and pH), hematological parameters (basophils, leukocytes, eosinophils, erythrocytes mean corpuscular hemoglobin, erythrocytes, hematocrit, hemoglobin, lymphocytes, mean platelet volume, monocytes, neutrophils, and platelets), and blood chemistry parameters (alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, calcium, chloride, cholesterol, creatinine, gamma glutamyl transferase, glucose, cholesterol, phosphate, potassium, protein, sodium, triglycerides, and urea nitrogen). Any laboratory result outside of the testing laboratory's normal range was classified as "clinically significant" or "not clinically significant" by the site investigator, with appropriate documentation.
Time Frame: Day 28
Population: SAS. Only participants with at least one clinically significant abnormal laboratory finding are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 42 | 19 | 23 | 13 | 41 | 43
Participants
  Urine occult blood - abnormal, clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Urine protein - abnormal, clinically significant | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Urine specimen appearance - abnormal, clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

35. Secondary Outcome: GMTs of HI Antibody Response for Each Homologous Influenza Strain on Day 182 and Day 365
Description: as for outcome 1
Time Frame: Day 182, Day 365
Population: Participants in PP Set with available data at each time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 37 | 18 | 21 | 13 | 34 | 33
titers
  H1N1: Day 182 | 226.2152 [133.2240 to 384.1147] | 332.5919 [154.1053 to 717.8036] | 175.6786 [120.2111 to 256.7397] | 129.4173 [75.1194 to 222.9628] | 118.8437 [71.8225 to 196.6492] | 214.5054 [113.0981 to 406.8378] | 164.9504 [111.0359 to 245.0435] | 121.7951 [81.4995 to 182.0140]
  H1N1: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  H1N1: Day 365 | 145.2654 [84.0127 to 251.1768] | 160.1136 [73.8080 to 347.3383] | 97.7443 [64.3983 to 148.3572] | 103.0787 [56.5787 to 187.7954] | 109.2066 [64.9584 to 183.5956] | 156.0724 [81.9383 to 297.2795] | 124.5817 [82.6212 to 187.8527] | 79.1142 [52.1240 to 120.0802]
  H3N2: Day 182 | 119.5465 [62.8739 to 227.3021] | 153.9351 [60.5150 to 391.5723] | 178.9880 [112.9393 to 283.6629] | 129.5061 [66.9232 to 250.6131] | 99.1267 [53.7954 to 182.6569] | 220.4298 [101.3667 to 479.3418] | 219.2384 [135.6131 to 354.4308] | 131.0605 [80.4859 to 213.4146]
  H3N2: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  H3N2: Day 365 | 156.9806 [81.6759 to 301.7156] | 217.4477 [86.3116 to 547.8233] | 189.1376 [114.9632 to 311.1694] | 210.9250 [103.1083 to 431.4819] | 141.6148 [76.1935 to 263.2082] | 265.6521 [123.1469 to 573.0639] | 254.8805 [156.1431 to 416.0547] | 135.1917 [82.1734 to 222.4177]
  B/Yamagata lineage: Day 182 | 45.3843 [25.4806 to 80.8353] | 83.0475 [35.8984 to 192.1226] | 50.0023 [33.0630 to 75.6203] | 33.5742 [18.5541 to 60.7534] | 30.1800 [17.4285 to 52.2611] | 33.1521 [16.4982 to 66.6173] | 46.0555 [29.9140 to 70.9067] | 51.3900 [33.1630 to 79.6348]
  B/Yamagata lineage: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  B/Yamagata lineage: Day 365 | 38.5246 [21.3868 to 69.3952] | 65.9800 [28.7046 to 151.6606] | 32.2612 [20.6025 to 50.5174] | 34.7689 [18.2475 to 66.2486] | 30.8130 [17.6303 to 53.8529] | 24.0753 [12.0453 to 48.1200] | 45.4888 [29.2558 to 70.7291] | 45.1481 [28.8323 to 70.6969]
  B/Victoria lineage: Day 182 | 33.2709 [20.3499 to 54.3959] | 44.8356 [21.9488 to 91.5873] | 59.2611 [41.6653 to 84.2879] | 39.9246 [24.0928 to 66.1598] | 42.7246 [26.7668 to 68.1960] | 52.2104 [28.8168 to 94.5952] | 37.2192 [25.7730 to 53.7489] | 43.4396 [29.9146 to 63.0796]
  B/Victoria lineage: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  B/Victoria lineage: Day 365 | 40.6922 [24.4797 to 67.6421] | 44.9239 [21.8954 to 92.1727] | 55.2532 [37.5128 to 81.3833] | 31.7135 [18.1750 to 55.3369] | 39.9398 [24.6619 to 64.6823] | 50.8227 [27.9482 to 92.4190] | 49.0601 [33.5119 to 71.8221] | 39.9694 [27.1362 to 58.8715]

36. Secondary Outcome: Percentage of Participants With Seroconversion Measured by HI Antibody Response for Each Homologous Influenza Strain on Day 182 and Day 365
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥4-fold increase in reciprocal HI titers between Day 0 and Day 182 and Day 0 and Day 365 or a rise of undetectable HI titer (i.e. <10) pre-vaccination (Day 0) to an HI titer of ≥40 on Day 182 and Day 365 was measured using an HI assay for the following homologous influenza strains: A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination) up to Day 182 and up to Day 365
Population: Participants in PP Set with available data at each timepoint were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 37 | 18 | 21 | 13 | 34 | 33
percentage of participants
  H1N1: Day 182 | 36.8 [16.29 to 61.64] | 55.6 [21.20 to 86.30] | 16.2 [6.19 to 32.01] | 27.8 [9.69 to 53.48] | 28.6 [11.28 to 52.18] | 38.5 [13.86 to 68.42] | 29.4 [15.10 to 47.48] | 27.3 [13.30 to 45.52]
  H1N1: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  H1N1: Day 365 | 27.8 [9.69 to 53.48] | 33.3 [7.49 to 70.07] | 22.6 [9.59 to 41.10] | 26.7 [7.79 to 55.10] | 25.0 [8.66 to 49.10] | 38.5 [13.86 to 68.42] | 12.5 [3.51 to 28.99] | 12.9 [3.63 to 29.83]
  H3N2: Day 182 | 31.6 [12.58 to 56.55] | 55.6 [21.20 to 86.30] | 32.4 [18.01 to 49.79] | 50.0 [26.02 to 73.98] | 42.9 [21.82 to 65.98] | 38.5 [13.86 to 68.42] | 47.1 [29.78 to 64.87] | 45.5 [28.11 to 63.65]
  H3N2: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  H3N2: Day 365 | 38.9 [17.30 to 64.25] | 44.4 [13.70 to 78.80] | 38.7 [21.85 to 57.81] | 46.7 [21.27 to 73.41] | 60.0 [36.05 to 80.88] | 61.5 [31.58 to 86.14] | 53.1 [34.74 to 70.91] | 45.2 [27.32 to 63.97]
  B/Yamagata lineage: Day 182 | 15.8 [3.38 to 39.58] | 11.1 [0.28 to 48.25] | 13.5 [4.54 to 28.77] | 0 [0.00 to 18.53] | 9.5 [1.17 to 30.38] | 7.7 [0.19 to 36.03] | 17.6 [6.76 to 34.53] | 24.2 [11.09 to 42.26]
  B/Yamagata lineage: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  B/Yamagata lineage: Day 365 | 11.1 [1.38 to 34.71] | 11.1 [0.28 to 48.25] | 9.7 [2.04 to 25.75] | 6.7 [0.17 to 31.95] | 15.0 [3.21 to 37.89] | 0 [0.00 to 24.71] | 3.1 [0.08 to 16.22] | 19.4 [7.45 to 37.47]
  B/Victoria lineage: Day 182 | 5.3 [0.13 to 26.03] | 22.2 [2.81 to 60.01] | 13.5 [4.54 to 28.77] | 22.2 [6.41 to 47.64] | 19.0 [5.45 to 41.91] | 0 [0.00 to 24.71] | 5.9 [0.72 to 19.68] | 21.2 [8.98 to 38.91]
  B/Victoria lineage: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  B/Victoria lineage: Day 365 | 5.6 [0.14 to 27.29] | 22.2 [2.81 to 60.01] | 9.7 [2.04 to 25.75] | 20.0 [4.33 to 48.09] | 5.0 [0.13 to 24.87] | 0 [0.00 to 24.71] | 3.1 [0.08 to 16.22] | 16.1 [5.45 to 33.73]

37. Secondary Outcome: Percentage of Participants With Seroprotection Measured by HI Antibody Response for Each Homologous Influenza Strain on Day 182 and Day 365
Description: Seroprotection rate: the percentage of participants in a given treatment group attaining a reciprocal HI titer of ≥40 on Day 182 and on Day 365 (the percentage of vaccine recipients with a serum HI titer of at least 1:40 following vaccination) for the homologous influenza strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage)
Time Frame: Day 0 (pre-vaccination) up to Day 182 and up to Day 365
Population: Participants in PP Set with available data at each timepoint were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 37 | 18 | 21 | 13 | 34 | 33
percentage of participants
  H1N1: Day 182 | 100 [82.35 to 100.00] | 100 [66.37 to 100.00] | 94.6 [81.81 to 99.34] | 94.4 [72.71 to 99.86] | 81.0 [58.09 to 94.55] | 100 [75.29 to 100.00] | 94.1 [80.32 to 99.28] | 97.0 [84.24 to 99.92]
  H1N1: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  H1N1: Day 365 | 27.8 [9.69 to 53.48] | 33.3 [7.49 to 70.07] | 22.6 [9.59 to 41.10] | 26.7 [7.79 to 55.10] | 25.0 [8.66 to 49.10] | 38.5 [13.86 to 68.42] | 12.5 [3.51 to 28.99] | 12.9 [3.63 to 29.83]
  H3N2: Day 182 | 89.5 [66.86 to 98.70] | 88.9 [51.75 to 99.72] | 94.6 [81.81 to 99.34] | 83.3 [58.58 to 96.42] | 90.5 [69.62 to 98.83] | 100 [75.29 to 100.00] | 91.2 [76.32 to 98.14] | 84.8 [68.10 to 94.89]
  H3N2: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  H3N2: Day 365 | 38.9 [17.30 to 64.25] | 44.4 [13.70 to 78.80] | 38.7 [21.85 to 57.81] | 46.7 [21.27 to 73.41] | 60.0 [36.05 to 80.88] | 61.5 [31.58 to 86.14] | 53.1 [34.74 to 70.91] | 45.2 [27.32 to 63.97]
  B/Yamagata lineage: Day 182 | 57.9 [33.50 to 79.75] | 88.9 [51.75 to 99.72] | 62.2 [44.76 to 77.54] | 50.0 [26.02 to 73.98] | 38.1 [18.11 to 61.56] | 46.2 [19.22 to 74.87] | 58.8 [40.70 to 75.35] | 69.7 [51.29 to 84.41]
  B/Yamagata lineage: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  B/Yamagata lineage: Day 365 | 11.1 [1.38 to 34.71] | 11.1 [0.28 to 48.25] | 9.7 [2.04 to 25.75] | 6.7 [0.17 to 31.95] | 15.0 [3.21 to 37.89] | 0 [0.00 to 24.71] | 3.1 [0.08 to 16.22] | 19.4 [7.45 to 37.47]
  B/Victoria lineage: Day 182 | 47.4 [24.45 to 71.14] | 77.8 [39.99 to 97.19] | 75.7 [58.80 to 88.23] | 50.0 [26.02 to 73.98] | 66.7 [43.03 to 85.41] | 69.2 [38.57 to 90.91] | 61.8 [43.56 to 77.83] | 66.7 [48.17 to 82.04]
  B/Victoria lineage: Day 365: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  B/Victoria lineage: Day 365 | 5.6 [0.14 to 27.29] | 22.2 [2.81 to 60.01] | 9.7 [2.04 to 25.75] | 20.0 [4.33 to 48.09] | 5.0 [0.13 to 24.87] | 0 [0.00 to 24.71] | 3.1 [0.08 to 16.22] | 16.1 [5.45 to 33.73]

38. Secondary Outcome: GMFR Measured by HI Antibody Response for Each Homologous Influenza Strain (Day 182/Day 0 and Day 365/Day 0)
Description: GMFR: the geometric mean of the ratio of GMTs (Day 182/Day 0 and Day 365/Day 0) measured using an HI assay for the homologous strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination), Day 182, Day 365
Population: Participants in PP Set with available data at each timepoint were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 37 | 18 | 21 | 13 | 34 | 33
ratio
  H1N1: Day 182/Day 0 | 2.8586 [1.7764 to 4.5999] | 4.6671 [2.3416 to 9.3021] | 2.4366 [1.7340 to 3.4239] | 1.9075 [1.1710 to 3.1072] | 1.7392 [1.1071 to 2.7322] | 1.9829 [1.9829 to 6.2724] | 2.1950 [1.5387 to 3.1310] | 1.7267 [1.2044 to 2.4754]
  H1N1: Day 365/Day 0: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  H1N1: Day 365/Day 0 | 1.7840 [1.1381 to 2.7964] | 2.2667 [1.2027 to 4.2720] | 1.6031 [1.1380 to 2.2583] | 1.6790 [1.0269 to 2.7451] | 1.6075 [1.0508 to 2.4592] | 2.7253 [1.6057 to 4.6254] | 1.5400 [1.0986 to 2.1588] | 1.1081 [0.7875 to 1.5593]
  H3N2: Day 182/Day 0 | 2.7326 [1.5003 to 4.9771] | 3.7625 [1.5737 to 8.9954] | 3.7985 [2.4701 to 5.8414] | 3.6059 [1.9379 to 6.7095] | 2.6792 [1.5087 to 4.7577] | 4.5291 [2.1919 to 9.3586] | 4.6788 [2.9870 to 7.3287] | 2.7380 [1.7355 to 4.3198]
  H3N2: Day 365/Day 0: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  H3N2: Day 365/Day 0 | 3.5029 [1.9348 to 6.3418] | 5.3618 [2.3150 to 12.4188] | 4.0557 [2.5792 to 6.3774] | 5.5988 [2.9159 to 10.7504] | 4.0497 [2.2937 to 7.1501] | 5.3933 [2.6799 to 10.8540] | 5.2951 [3.3896 to 8.2719] | 2.8866 [1.8356 to 4.5393]
  B/Yamagata lineage: Day 182/Day 0 | 1.5914 [1.0554 to 2.3995] | 1.8261 [1.0027 to 3.3256] | 1.4557 [1.0841 to 1.9546] | 1.2508 [0.8200 to 1.9080] | 1.1448 [0.7742 to 1.6928] | 2.2374 [0.8272 to 2.2374] | 1.5232 [1.1206 to 2.0704] | 1.5720 [1.1511 to 2.1470]
  B/Yamagata lineage: Day 365/Day 0: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  B/Yamagata lineage: Day 365/Day 0 | 1.3110 [0.8696 to 1.9765] | 1.4345 [0.8000 to 2.5722] | 1.1944 [0.8731 to 1.6338] | 1.2518 [0.7983 to 1.9630] | 1.1462 [0.7761 to 1.6926] | 0.9986 [0.6153 to 1.6207] | 1.3226 [0.9716 to 1.8005] | 1.3422 [0.9813 to 1.8358]
  B/Victoria lineage: Day 182/Day 0 | 0.9854 [0.6970 to 1.3930] | 1.2056 [0.7291 to 1.9937] | 1.3892 [1.0824 to 1.7830] | 1.4917 [1.0429 to 2.1338] | 1.1803 [0.8492 to 1.6405] | 1.0689 [0.7015 to 1.6287] | 1.1041 [0.8523 to 1.4303] | 1.4098 [1.0833 to 1.8346]
  B/Victoria lineage: Day 365/Day 0: number analyzed (Participants) | 18 | 9 | 31 | 15 | 20 | 13 | 32 | 31
  B/Victoria lineage: Day 365/Day 0 | 1.1788 [0.8363 to 1.6615] | 1.1979 [0.7372 to 1.9463] | 1.3199 [1.0153 to 1.7159] | 1.2063 [0.8261 to 1.7615] | 1.1095 [0.8012 to 1.5365] | 1.0238 [0.6819 to 1.5371] | 1.2542 [0.9693 to 1.6229] | 1.3656 [1.0496 to 1.7767]

39. Secondary Outcome: GMTs of HI Antibody Response for Each Heterologous Influenza Strain
Description: The GMTs in each treatment group were measured using an HI assay for the heterologous influenza strains: A/Brisbane/02/2018 (H1N1), A/Kansas/14/2017 (H3N2), and B/Maryland/15/2016 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination), Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 38 | 19 | 21 | 13 | 37 | 39
titers
  H1N1: Day 0 | 90.8941 [46.5459 to 177.4963] | 60.8920 [23.0277 to 161.0166] | 57.0448 [35.5380 to 91.5672] | 29.8495 [15.2856 to 58.2896] | 45.6156 [24.1349 to 86.2145] | 35.0221 [15.5941 to 78.6549] | 58.6793 [36.3248 to 94.7911] | 36.2950 [22.7497 to 57.9053]
  H1N1: Day 28: number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
  H1N1: Day 28 | 290.5308 [152.0669 to 555.0723] | 418.9367 [167.6995 to 1046.5621] | 191.9608 [122.9439 to 299.7219] | 90.8596 [48.3851 to 170.6197] | 107.3121 [58.0657 to 198.3253] | 168.6130 [78.7144 to 361.1836] | 141.5521 [88.3780 to 226.7192] | 210.6752 [135.7077 to 327.0561]
  H3N2: Day 0 | 38.5796 [20.3087 to 73.2878] | 21.6012 [8.5030 to 54.8760] | 32.0958 [20.3890 to 50.5243] | 17.5909 [9.2601 to 33.4167] | 16.9318 [9.1967 to 31.1729] | 30.5442 [14.0614 to 66.3484] | 40.3477 [25.4754 to 63.9023] | 25.6289 [16.3764 to 40.1088]
  H3N2: Day 28: number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
  H3N2: Day 28 | 89.5835 [45.8327 to 175.0980] | 56.5609 [21.9233 to 145.9243] | 79.9144 [50.3858 to 126.7481] | 47.9629 [24.9813 to 92.0864] | 36.6176 [19.3898 to 69.1524] | 48.0514 [21.8386 to 105.7274] | 108.5069 [66.6323 to 176.6971] | 121.5473 [77.0928 to 191.6358]
  B/Victoria lineage: Day 0 | 22.6953 [12.6605 to 40.6840] | 38.4838 [16.4805 to 89.8640] | 34.2028 [22.6370 to 51.6779] | 14.9040 [8.3141 to 26.7171] | 18.0797 [10.3771 to 31.4995] | 18.4484 [9.1098 to 37.3602] | 26.9646 [17.7478 to 40.9677] | 14.8765 [9.8986 to 22.3579]
  B/Victoria lineage: Day 28: number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
  B/Victoria lineage: Day 28 | 39.2478 [22.4411 to 68.6416] | 58.8887 [26.7117 to 129.8263] | 65.9266 [44.8718 to 96.8606] | 22.2497 [12.9130 to 38.3371] | 31.8255 [18.7268 to 54.0865] | 27.5162 [14.2535 to 53.1199] | 45.6899 [30.4213 to 68.6218] | 59.6513 [40.8027 to 87.2069]

40. Secondary Outcome: Percentage of Participants With Seroconversion Measured by HI Antibody Response for Each Heterologous Influenza Strain
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥4-fold increase in reciprocal HI titers between Day 0 and Day 28 or a rise of undetectable HI titer (i.e. <10) pre-vaccination (Day 0) to an HI titer of ≥40 on Day 28 was measured using an HI assay for the heterologous influenza strains A/Brisbane/02/2018 (H1N1), A/Kansas/14/2017 (H3N2), and B/Maryland/15/2016 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
percentage of participants
  H1N1 | 33.3 [13.34 to 59.01] | 55.6 [21.20 to 86.30] | 36.8 [21.81 to 54.01] | 31.6 [12.58 to 56.55] | 25.0 [8.66 to 49.10] | 38.5 [13.86 to 68.42] | 29.4 [15.10 to 47.48] | 53.8 [37.18 to 69.91]
  H3N2 | 16.7 [3.58 to 41.42] | 33.3 [7.49 to 70.07] | 18.4 [7.74 to 34.33] | 26.3 [9.15 to 51.20] | 20.0 [5.73 to 43.66] | 15.4 [1.92 to 45.45] | 29.4 [15.10 to 47.48] | 53.8 [37.18 to 69.91]
  B/Victoria lineage | 11.1 [1.38 to 34.71] | 11.1 [0.28 to 48.25] | 13.2 [4.41 to 28.09] | 5.3 [0.13 to 26.03] | 15.0 [3.21 to 37.89] | 7.7 [0.19 to 36.03] | 11.8 [3.30 to 27.45] | 46.2 [30.09 to 62.82]

41. Secondary Outcome: Percentage of Participants With Seroprotection Measured by HI Antibody Response for Each Heterologous Influenza Strain
Description: Seroprotection rate: the percentage of participants in a given treatment group attaining a reciprocal HI titer of ≥40 on Day 28 (the percentage of vaccine recipients with a serum HI titer of at least 1:40 following vaccination) for the heterologous influenza strains A/Brisbane/02/2018 (H1N1), A/Kansas/14/2017 (H3N2), and B/Maryland/15/2016 (B/Victoria lineage)
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 38 | 19 | 20 | 13 | 34 | 39
percentage of participants
  H1N1: number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
  H1N1 | 100 [81.47 to 100.00] | 100 [66.37 to 100.00] | 89.5 [75.20 to 97.06] | 78.9 [54.43 to 93.95] | 80.0 [56.34 to 94.27] | 84.6 [54.55 to 98.08] | 88.2 [72.55 to 96.70] | 92.3 [79.13 to 98.38]
  H3N2: number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
  H3N2 | 72.2 [46.52 to 90.31] | 66.7 [29.93 to 92.51] | 73.7 [56.90 to 86.60] | 57.9 [33.50 to 79.75] | 55.0 [31.53 to 76.94] | 53.8 [25.13 to 80.78] | 79.4 [62.10 to 91.30] | 89.7 [75.78 to 97.13]
  B/Victoria lineage: number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
  B/Victoria lineage | 61.1 [35.75 to 82.70] | 77.8 [39.99 to 97.19] | 71.1 [54.10 to 84.58] | 42.1 [20.25 to 66.50] | 45.0 [23.06 to 68.47] | 61.5 [31.58 to 86.14] | 64.7 [46.49 to 80.25] | 76.9 [60.67 to 88.87]

42. Secondary Outcome: GMFR Measured by HI Antibody Response for Each Heterologous Influenza Strain
Description: GMFR: the geometric mean of the ratio of GMTs (Day 28/Day 0) measured using an HI assay for the heterologous strains A/Brisbane/02/2018 (H1N1), A/Kansas/14/2017 (H3N2), and B/Maryland/15/2016 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination), Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 18 | 9 | 38 | 19 | 20 | 13 | 34 | 39
ratio
  H1N1 | 4.6104 [2.6534 to 8.0105] | 7.7661 [3.5725 to 16.8825] | 3.6764 [2.5186 to 5.3663] | 2.4044 [1.4056 to 4.1130] | 2.2511 [1.3376 to 3.7885] | 4.1198 [2.1579 to 7.8655] | 2.7513 [1.8449 to 4.1028] | 5.0566 [3.4783 to 7.3510]
  H3N2 | 2.8906 [1.6272 to 5.1350] | 2.3315 [1.0348 to 5.2531] | 2.6710 [1.7985 to 3.9667] | 2.2043 [1.2571 to 3.8651] | 1.7248 [0.9969 to 2.9842] | 1.6487 [0.8391 to 3.2397] | 3.2113 [2.1092 to 4.8895] | 4.5766 [3.0985 to 6.7598]
  B/Victoria lineage | 1.7604 [1.1839 to 2.6177] | 1.8557 [1.0562 to 3.2605] | 2.2441 [1.7023 to 2.9582] | 1.3040 [0.8847 to 1.9221] | 1.6675 [1.1438 to 2.4310] | 1.4026 [0.8791 to 2.2377] | 1.7975 [1.3458 to 2.4008] | 3.5002 [2.6662 to 4.5950]

43. Secondary Outcome: GMTs of Microneutralization (MN) Antibody Response for Each Homologous Influenza Strain
Description: The GMTs in each treatment group were measured using an MN assay for the homologous influenza strains: A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination), Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 19 | 9 | 38 | 19 | 21 | 13 | 36 | 38
titers
  H1N1: Day 0: number analyzed (Participants) | 19 | 8 | 38 | 18 | 21 | 13 | 36 | 38
  H1N1: Day 0 | 195.2871 [96.6328 to 394.6597] | 216.6401 [73.2581 to 640.6514] | 127.4353 [77.4879 to 209.5779] | 137.0522 [66.5218 to 282.3630] | 122.6834 [62.8276 to 239.5636] | 93.8593 [40.0947 to 219.7194] | 141.0830 [84.6249 to 235.2074] | 89.1100 [54.1840 to 146.5489]
  H1N1: Day 28: number analyzed (Participants) | 18 | 9 | 38 | 19 | 19 | 13 | 34 | 38
  H1N1: Day 28 | 887.6906 [435.2611 to 1810.3950] | 1956.7218 [714.1894 to 5360.9873] | 663.8670 [406.4999 to 1084.1807] | 495.8821 [247.8117 to 992.2818] | 532.9893 [266.3556 to 1066.5349] | 693.3781 [299.7565 to 1603.8791] | 434.8282 [258.8898 to 730.3325] | 754.0606 [461.7274 to 1231.4786]
  H3N2: Day 0: number analyzed (Participants) | 19 | 7 | 38 | 18 | 21 | 13 | 36 | 38
  H3N2: Day 0 | 123.9489 [82.3861 to 186.4795] | 107.6687 [54.9339 to 211.0273] | 96.9336 [72.6176 to 129.3919] | 84.7454 [55.7015 to 128.9334] | 65.5761 [44.4647 to 96.7110] | 129.3964 [78.9714 to 212.0188] | 98.8487 [73.4685 to 132.9967] | 100.5515 [75.3279 to 134.2212]
  H3N2: Day 28: number analyzed (Participants) | 16 | 9 | 32 | 16 | 19 | 10 | 30 | 35
  H3N2: Day 28 | 198.6618 [139.6367 to 282.6371] | 332.5998 [207.8591 to 532.2001] | 205.2176 [159.9359 to 263.3195] | 186.1487 [130.8414 to 264.8346] | 188.4193 [136.3382 to 260.3952] | 196.9789 [126.1081 to 307.6778] | 216.0005 [166.9689 to 279.4306] | 273.0912 [215.1708 to 346.6029]
  B/Yamagata lineage: Day 0: number analyzed (Participants) | 17 | 8 | 33 | 15 | 20 | 13 | 33 | 37
  B/Yamagata lineage: Day 0 | 16.3090 [9.8086 to 27.1173] | 17.5404 [8.3588 to 36.8073] | 18.9617 [13.1640 to 27.3129] | 10.7232 [6.2408 to 18.4248] | 10.8996 [6.8206 to 17.4178] | 10.2622 [5.7375 to 18.3551] | 20.6308 [14.3227 to 29.7171] | 22.3655 [15.8453 to 31.5688]
  B/Yamagata lineage: Day 28: number analyzed (Participants) | 15 | 9 | 29 | 15 | 18 | 13 | 27 | 30
  B/Yamagata lineage: Day 28 | 25.7962 [15.8706 to 41.9293] | 34.2802 [18.3102 to 64.1793] | 38.0649 [26.8412 to 53.9819] | 15.4893 [9.5295 to 25.1765] | 21.5952 [13.8604 to 33.6464] | 15.7214 [9.3300 to 26.4911] | 30.5144 [21.2453 to 43.8276] | 64.2153 [45.5476 to 90.5340]
  B/Victoria lineage: Day 0: number analyzed (Participants) | 19 | 8 | 38 | 18 | 21 | 13 | 36 | 38
  B/Victoria lineage: Day 0 | 25.7760 [14.6760 to 45.2712] | 25.9287 [10.8847 to 61.7654] | 34.8450 [23.3979 to 51.8924] | 15.8462 [8.8842 to 28.2642] | 15.3550 [8.9863 to 26.2372] | 29.8305 [15.0989 to 58.9354] | 22.2014 [14.7461 to 33.4260] | 14.2585 [9.5743 to 21.2342]
  B/Victoria lineage: Day 28: number analyzed (Participants) | 18 | 9 | 37 | 18 | 19 | 13 | 34 | 38
  B/Victoria lineage: Day 28 | 42.3874 [22.1575 to 81.0874] | 104.7367 [41.8496 to 262.1236] | 70.2059 [44.6561 to 110.3740] | 36.2627 [18.9559 to 69.3709] | 45.4444 [24.1700 to 85.4443] | 75.8887 [35.3738 to 162.8065] | 33.2720 [20.7539 to 53.3406] | 64.2444 [41.1098 to 100.3983]

44. Secondary Outcome: Percentage of Participants With Seroconversion Measured by MN Antibody Response for Each Homologous Influenza Strain
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥4-fold increase in reciprocal HI titers between Day 0 and Day 28 or a rise of undetectable MN titer (i.e. <10) pre-vaccination (Day 0) to an MN titer of ≥40 on Day 28 was measured using an MN assay for the homologous influenza strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 18 | 8 | 38 | 18 | 19 | 13 | 33 | 37
percentage of participants
  H1N1 | 38.9 [17.30 to 64.25] | 50.0 [15.70 to 84.30] | 55.3 [38.30 to 71.38] | 33.3 [13.34 to 59.01] | 42.1 [20.25 to 66.50] | 61.5 [31.58 to 86.14] | 33.3 [17.96 to 51.83] | 59.5 [42.10 to 75.25]
  H3N2: number analyzed (Participants) | 16 | 7 | 32 | 15 | 19 | 10 | 29 | 34
  H3N2 | 12.5 [1.55 to 38.35] | 42.9 [9.90 to 81.59] | 15.6 [5.28 to 32.79] | 26.7 [7.79 to 55.10] | 42.1 [20.25 to 66.50] | 10.0 [0.25 to 44.50] | 17.2 [5.85 to 35.77] | 35.3 [19.75 to 53.51]
  B/Yamagata lineage: number analyzed (Participants) | 15 | 8 | 29 | 14 | 18 | 13 | 26 | 29
  B/Yamagata lineage | 20.0 [4.33 to 48.09] | 12.5 [0.32 to 52.65] | 17.2 [5.85 to 35.77] | 7.1 [0.18 to 33.87] | 22.2 [6.41 to 47.64] | 0 [0.00 to 24.71] | 3.8 [0.10 to 19.64] | 34.5 [17.94 to 54.33]
  B/Victoria lineage: number analyzed (Participants) | 18 | 8 | 37 | 17 | 19 | 13 | 33 | 37
  B/Victoria lineage | 5.6 [0.14 to 27.29] | 25.0 [3.19 to 65.09] | 18.9 [7.96 to 35.16] | 29.4 [10.31 to 55.96] | 26.3 [9.15 to 51.20] | 30.8 [9.09 to 61.43] | 15.2 [5.11 to 31.90] | 43.2 [27.10 to 60.51]

45. Secondary Outcome: GMFR Measured by MN Antibody Response for Each Homologous Influenza Strain
Description: GMFR: the geometric mean of the ratio of GMTs (Day 28/Day 0) measured using an MN assay for the homologous strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage).
Time Frame: Day 0 (pre-vaccination), Day 28
Population: Participants in PP Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 18 | 8 | 38 | 18 | 19 | 13 | 33 | 37
ratio
  H1N1 | 6.0914 [3.2359 to 11.4669] | 12.7121 [4.9188 to 32.8531] | 5.2592 [3.4061 to 8.1206] | 4.0415 [2.1497 to 7.5982] | 4.0654 [2.1990 to 7.5158] | 6.3495 [3.0183 to 13.3571] | 3.4096 [2.1392 to 5.4344] | 6.5345 [4.2010 to 10.1641]
  H3N2: number analyzed (Participants) | 16 | 7 | 32 | 15 | 19 | 10 | 29 | 34
  H3N2 | 1.8781 [1.3659 to 2.5824] | 2.7393 [1.6952 to 4.4264] | 2.1798 [1.7414 to 2.7287] | 2.0133 [1.4499 to 2.7956] | 2.1935 [1.6353 to 2.9422] | 1.8735 [1.2531 to 2.8010] | 2.1377 [1.6879 to 2.7074] | 2.8084 [2.2590 to 3.4914]
  B/Yamagata lineage: number analyzed (Participants) | 15 | 8 | 29 | 14 | 18 | 13 | 26 | 29
  B/Yamagata lineage | 1.7366 [1.1767 to 2.5629] | 1.8812 [1.1036 to 3.2068] | 2.3239 [1.7552 to 3.0767] | 1.3802 [0.9177 to 2.0758] | 1.7651 [1.2341 to 2.5247] | 1.3086 [0.8592 to 1.9930] | 1.8310 [1.3613 to 2.4628] | 3.5437 [2.6727 to 4.6986]
  B/Victoria lineage: number analyzed (Participants) | 18 | 8 | 37 | 17 | 19 | 13 | 33 | 37
  B/Victoria lineage | 1.7152 [1.0254 to 2.8691] | 4.4083 [2.0388 to 9.5320] | 2.4424 [1.7000 to 3.5091] | 2.3549 [1.3853 to 4.0032] | 2.4501 [1.4844 to 4.0440] | 2.8024 [1.5286 to 5.1377] | 1.5535 [1.0629 to 2.2706] | 3.8216 [2.6602 to 5.4898]

46. Secondary Outcome: GMTs of HI Antibody Response for Each Homologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: The GMTs in each treatment group were measured using an HI assay for the homologous influenza strains: A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination), Day 28
Population: The analysis was not performed because less than 25% of the enrolled participants had received a standard influenza vaccine during the last 12 months prior to study vaccination.
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Percentage of Participants With Seroconversion Measured by HI Antibody Response for Each Homologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥4-fold increase in reciprocal HI titers between Day 0 and Day 28 or a rise of undetectable HI titer (i.e. <10) pre-vaccination (Day 0) to an HI titer of ≥40 on Day 28 was measured using an HI assay for the homologous influenza strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

48. Secondary Outcome: Percentage of Participants With Seroprotection Measured by HI Antibody Response for Each Homologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: Seroprotection rate: the percentage of participants in a given treatment group attaining a reciprocal HI titer of ≥40 on Day 28 (the percentage of vaccine recipients with a serum HI titer of at least 1:40 following vaccination) for the homologous influenza strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: GMFR Measured by HI Antibody Response for Each Homologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: GMFR: the geometric mean of the ratio of GMTs (Day 28/Day 0) measured using an HI assay for the homologous strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination), Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

50. Secondary Outcome: GMTs of HI Antibody Response for Each Heterologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: The GMTs in each treatment group were measured using an HI assay for the heterologous influenza strains: A/Brisbane/02/2018 (H1N1), A/Kansas/14/2017 (H3N2), and B/Maryland/15/2016 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination), Day 28
Population: The analysis were not performed because less than 25% of the enrolled participants had received a standard influenza vaccine during the last 12 months prior to study vaccination.
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

51. Secondary Outcome: Percentage of Participants With Seroconversion Measured by HI Antibody Response for Each Heterologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥4-fold increase in reciprocal HI titers between Day 0 and Day 28 or a rise of undetectable HI titer (i.e. <10) pre-vaccination (Day 0) to an HI titer of ≥40 on Day 28 was measured using an HI assay for the following heterologous influenza strains: A/Brisbane/02/2018 (H1N1), A/Kansas/14/2017 (H3N2), and B/Maryland/15/2016 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

52. Secondary Outcome: Percentage of Participants With Seroprotection Measured by HI Antibody Response for Each Heterologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: Seroprotection rate: the percentage of participants in a given treatment group attaining a reciprocal HI titer of ≥40 on Day 28 (the percentage of vaccine recipients with a serum HI titer of at least 1:40 following vaccination) for the following heterologous influenza strains: A/Brisbane/02/2018 (H1N1), A/Kansas/14/2017 (H3N2), and B/Maryland/15/2016 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

53. Secondary Outcome: GMFR Measured by HI Antibody Response for Each Heterologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: GMFR: the geometric mean of the ratio of GMTs (Day 28/Day 0) measured using an HI assay for the heterologous strains A/Brisbane/02/2018 (H1N1), A/Kansas/14/2017 (H3N2), and B/Maryland/15/2016 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination), Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

54. Secondary Outcome: GMTs of MN Antibody Response for Each Homologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: The GMTs in each treatment group were measured using an MN assay for the following homologous influenza strains: A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination), Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

55. Secondary Outcome: Percentage of Participants With Seroconversion Measured by MN Antibody Response for Each Homologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥4-fold increase in reciprocal HI titers between Day 0 and Day 28 or a rise of undetectable MN titer (i.e. <10) pre-vaccination (Day 0) to an MN titer of ≥40 on Day 28 was measured using an MN assay for the homologous influenza strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

56. Secondary Outcome: GMFR Measured by MN Antibody Response for Each Homologous Influenza Strain, Stratified by Prior Influenza Vaccination Status
Description: GMFR: the geometric mean of the ratio of GMTs (Day 28/Day 0) measured using an MN assay for the strains A/Hawaii/70/2019 (H1N1), A/Minnesota/41/2019 (H3N2), B/Singapore/INFKK-16-0569/2016 (B/Yamagata lineage), and B/Washington/02/2019 (B/Victoria lineage). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination), Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Number of Participants With at Least One Immediate AE, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. Immediate AEs were defined as any solicited (local and systemic) and unsolicited AEs that started up to 30 minutes after vaccination. Solicited local AEs included erythema, swelling and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Up to 30 minutes post-vaccination
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

58. Secondary Outcome: Number of Participants With at Least One Immediate AE of Grade 1, 2, 3, or 4, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined in OM #6. Immediate AEs were defined as any solicited (local and systemic) and unsolicited AEs that started up to 30 minutes after vaccination. Solicited local AEs included erythema, swelling and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck. The intensity of the AEs was graded according to the FDA Toxicity Grading Scale: mild (Grade 1), moderate (Grade 2), severe (Grade 3), or potentially life threatening (Grade 4). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Up to 30 minutes post-vaccination
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

59. Secondary Outcome: Number of Participants With at Least One Immediate AE Related to Vaccination, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined in OM #6. Immediate AEs were defined as any solicited (local and systemic) and unsolicited AEs that started up to 30 minutes after vaccination. Solicited local AEs included erythema, swelling and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck. A related AE is an event where the investigator determined that the relationship to study vaccine was "Possibly Related", "Probably Related", or "Definitely Related". If a participant reported multiple occurrences of the same AE, only the most closely related occurrence was presented. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Up to 30 minutes post-vaccination
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

60. Secondary Outcome: Number of Participants With at Least One Solicited Local or Systemic AE, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. Solicited local AEs included erythema, swelling and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 7
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

61. Secondary Outcome: Number of Participants With at Least One Solicited Local or Systemic AE of Grade 1, 2, 3, or 4, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. Solicited local AEs included erythema, swelling and pain at the injection site. Solicited systemic AEs included fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck. The intensity of the AEs was graded according to the FDA Toxicity Grading Scale: mild (Grade 1), moderate (Grade 2), severe (Grade 3), or potentially life threatening (Grade 4). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 7
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

62. Secondary Outcome: Number of Participants With at Least One Unsolicited AE, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

63. Secondary Outcome: Number of Participants With at Least One Unsolicited AE of Grade 1, 2, 3, or 4, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. The intensity of the AEs was graded according to the FDA Toxicity Grading Scale: mild (Grade 1), moderate (Grade 2), severe (Grade 3), or potentially life threatening (Grade 4). It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

64. Secondary Outcome: Number of Participants With at Least One Unsolicited AE Related to Vaccination, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. A related AE was an event where the Investigator determined that the relationship to study vaccine was "Possibly Related", "Probably Related", or "Definitely Related". It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination) up to Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

65. Secondary Outcome: Number of Participants With at Least One SAE From Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. An SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

66. Secondary Outcome: Number of Participants With at Least One AE Leading to Withdrawal From the Study From Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365, Stratified by Prior Influenza Vaccination Status
Description: as for outcome 62
Time Frame: Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

67. Secondary Outcome: Number of Participants With at Least One AESI From Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. AESIs included hypersensitivity reactions, narcolepsy, pIMDs, and other AESIs. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

68. Secondary Outcome: Number of Participants With at Least One MAAE From Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365, Stratified by Prior Influenza Vaccination Status
Description: An AE is defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. MAAEs are defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

69. Secondary Outcome: Number of Participants With at Least One NOCD From Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365, Stratified by Prior Influenza Vaccination Status
Description: All NOCDs that may plausibly have an allergic, autoimmune or inflammatory component were assessed and reported. Plausibility was interpreted broadly; the only clear exceptions were degenerative conditions such as osteoarthritis, age-related physiologic changes and life-style diseases. In this context, most cancers, cardiac conditions, and kidney diseases had to be reported. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

70. Secondary Outcome: Number of Participants With the Occurrence of Death From Day 1 up to Day 28, From Day 29 to Day 182, and From Day 183 to Day 365, Stratified by Prior Influenza Vaccination Status
Description: The number of participants in each treatment group with an occurrence of death was assessed. It was planned that the endpoint would be analyzed only if >25% of the enrolled participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 1 up to Day 28, Day 29 up to Day 182, and Day 183 up to Day 365
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

71. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Urine, Hematological, and Blood Biochemistry Values on Day 0, Stratified by Prior Influenza Vaccination Status
Description: Participants were monitored for abnormal findings in urine parameters (urine color, glucose, occult blood, protein, specific gravity, specimen appearance, pH), hematological parameters (basophils, leukocytes, eosinophils, erythrocytes mean corpuscular hemoglobin, erythrocytes, hematocrit, hemoglobin, lymphocytes, mean platelet volume, monocytes, neutrophils, platelets), and blood chemistry parameters (alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, calcium, chloride, cholesterol, creatinine, gamma glutamyl transferase, glucose, HDL and LDL cholesterol, phosphate, potassium, protein, sodium, triglycerides, urea nitrogen). Any laboratory result outside of the normal range was classified as "clinically significant" or "not clinically significant" by the site investigator. It was planned that the endpoint would be analyzed if >25% of the participants had received a standard influenza vaccine during the 12 months prior to study vaccination.
Time Frame: Day 0 (pre-vaccination)
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

72. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Urine, Hematological, and Blood Biochemistry Values on Day 3, Stratified by Prior Influenza Vaccination Status
Description: as for outcome 71
Time Frame: Day 3
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

73. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Urine, Hematological, and Blood Biochemistry Values on Day 28, Stratified by Prior Influenza Vaccination Status
Description: as for outcome 71
Time Frame: Day 28
Population: as for outcome 46
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 (post-vaccination) to Day 365 (end of study)
Description: SAS. The unsolicited SAEs, unsolicited non-serious AEs, and all deaths were reported.
Arm/Group | QVLP15+Full AS03 | QVLP15+Half AS03 | QVLP30+Full AS03 | QVLP30+Half AS03 | QVLP45+Full AS03 | QVLP45+Half AS03 | QVLP30 Unadjuvanted | Fluzone HD Quad
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/9 | 1/42 | 0/19 | 0/23 | 0/13 | 0/41 | 1/43
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/9 | 6/42 | 2/19 | 1/23 | 0/13 | 1/41 | 5/43
Other Adverse Events (participants affected / at risk) | 10/19 | 5/9 | 19/42 | 6/19 | 5/23 | 4/13 | 18/41 | 16/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVLP15+Full AS03 (N=19) | QVLP15+Half AS03 (N=9) | QVLP30+Full AS03 (N=42) | QVLP30+Half AS03 (N=19) | QVLP45+Full AS03 (N=23) | QVLP45+Half AS03 (N=13) | QVLP30 Unadjuvanted (N=41) | Fluzone HD Quad (N=43)
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVLP15+Full AS03 (N=19) | QVLP15+Half AS03 (N=9) | QVLP30+Full AS03 (N=42) | QVLP30+Half AS03 (N=19) | QVLP45+Full AS03 (N=23) | QVLP45+Half AS03 (N=13) | QVLP30 Unadjuvanted (N=41) | Fluzone HD Quad (N=43)
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Infection parasitic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 5 | 0 | 0 | 0 | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Perineal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator understands that the information in the protocol is confidential and should not be disclosed, other than to those directly involved in the execution or the ethical review of the study, without prior written authorization from the Sponsor. It is, however, permissible to discuss information contained in the protocol with a participant in order to obtain consent once Institutional Review Board (IRB) approval is obtained.

DOCUMENTS (2):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT04622592/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT04622592/SAP_001.pdf